CLINICAL TRIAL: NCT00178750
Title: A Randomized Clinical Comparison of the "Loss of Resistance" Technique Versus the CompuFlo® Computerized Syringe Pump for Proper Epidural Placement
Brief Title: "Loss of Resistance" Versus CompuFlo® for Epidural Placement
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study did not start due to investigator time constraints
Sponsor: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-04-248
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Pain; Epidural Analgesia
Keywords: Epidural placement; CompuFlo®
MeSH Terms: conditions — Pain

INTERVENTIONS:
Device: 18G Tuohy epidural needle
Device: CompuFlo® computerized syringe pump

SUMMARY:
The purpose of this study is to compare how well the CompuFlo® computerized syringe pump works as compared to the traditional method of inserting an epidural (a needle placed in one's back to give pain medicine).

DETAILED DESCRIPTION:
It is possible to utilize epidural anesthesia as the sole anesthetic technique for thoracic, abdominal, and lower extremity surgeries, as a method of postoperative pain management after surgery, and for pain relief during labor and delivery. However, despite the various benefits of epidural anesthesia, this procedure is not utilized to its maximum potential in the operating room. One reason for inadequate utilization of this procedure is the difficulty in properly identifying the epidural space. Current techniques for identifying the epidural space rely on the subjective perception of the operator on loss of resistance to air or saline as the needle passes from the ligamentum flavum into the epidural space. CompuFlo®'s pressure-sensing technology provides an objective measurement for proper placement of the epidural.

Very little advancement has been made in improving training to identify the correct location of the epidural space. Epidural anesthesia has a relatively higher failure rate when performed by residents in training. The skills of trainees differ greatly, and there are no standard teaching methods to teach epidural anesthesia. Statistical analysis conducted by Naik et al. concluded that some residents may need as many as 75 attempts at epidural anesthesia to ensure proficiency.

The CompuFlo® is a computerized syringe pump capable of volume and pressure-controlled infusion. It has a pressure sensor and a mathematical algorithm capable of determining the pressure at the needle tip. Pressures are continuously monitored and displayed, which are reflected by acoustic changes in tone. A dramatic pressure decrease and a high tissue compliance (pressure does not increase despite continuous infusion) signifies entrance into the epidural space. Combining a program with a low upper pressure limit and a high infusion rate mimics the technique used by the loss of resistance with saline proponents (constant pressure on the plunger). It combines the "feel" of inserting an epidural needle with the visualization of the pressure level, as well as a sound indicator to indicate proper placement.

ELIGIBILITY:
Inclusion Criteria:

* Any obstetric patient presenting for vaginal delivery desiring epidural anesthesia
* American Society of Anesthesiologists (ASA) Physical Classification I-III
* Aged 18-65 years

Exclusion Criteria:

* Obstetric patients presenting for Cesarean section
* American Society of Anesthesiologists Physical Classification ≥ IV
* Contraindications for epidural anesthesia
* Allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Number of attempts
Incidence of incorrect epidural placement
Pain level 1-10

SECONDARY OUTCOMES:
Subjective difficulty in placing epidural

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Ghelber, M.D., Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States